CLINICAL TRIAL: NCT01345448
Title: Study of Safety and IOP Lowering Efficacy of Transdermal Brimonidine Therapy
Brief Title: Intraocular Pressure (IOP) Lowering Efficacy of Transdermal Brimonidine Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanduri, Padma, M.D., FACS (Individual)
Responsible Party: Padma Nanduri, M.D., F.A.C.S., Padma Nanduri, M.D., F.A.C.S.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: White Rabbit 2010-0001
Record Dates: First submitted 2011-04-27; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Glaucoma
Keywords: Glaucoma; Brimonidine; Transdermal
MeSH Terms: conditions — Glaucoma | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Brimonidine — 0.1% Brimonidine Lotion, dosed once.
  Other Names: Alphagan
Drug: Placebo Lotion — Placebo Lotion dosed once.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness in lowering intraocular pressure (IOP) utilizing an experimental lotion containing 0.1% Brimonidine that is applied to the outside of one eyelid.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide, with primary open-angle glaucoma the most common form of glaucoma. Vision loss is caused by damage to the optic nerve. The modern goals of glaucoma management are to avoid glaucomatous damage, nerve damage, preserve visual field and total quality of life for patients with minimal side effects.

Although intraocular pressure is only one of the major risk factors for glaucoma, lowering it via various pharmaceuticals and/or surgical techniques is currently the mainstay of glaucoma treatment. Intraocular pressure can be lowered with medication, usually eye drops. There are several different classes of medications to treat glaucoma with several different medications in each class. In order to prevent blindness from glaucoma, it is critical that patients take their glaucoma eye drops accurately and faithfully for the rest of their lives. Poor compliance with medications and follow-up visits is a major reason for vision loss in glaucoma patients. In addition, coordination involved in placing an eye drop in the eye is considerably more difficult and unpleasant to patients than many other therapies. Thus, localized transdermal eyelid lotion would create a leap in safety of drug delivery while at the same time rendering ocular drugs easy and non traumatic to use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of stable Chronic Open Angle Glaucoma and stable Vital signs who are controlled on a stable dose of a single IOP lowering agent and who have demonstrated stable target intraocular pressure for a minimum of 3 months.
* Male or Female patients aged at least 18 years of age.
* Females of childbearing potential must use a reliable form of contraception throughout the study period such as celibacy, birth control pills, or condoms.
* A negative urine pregnancy test result at Screening and Baseline (Day 1) for women of childbearing potential
* Best-Corrected Visual Acuity of 20/800 or better in both eyes
* Written informed consent.
* Ability to follow instructions and likely to complete all study visits based upon patient factors such as cognition, reliability, motivation, and ability to obtain reliable transportation to study site.

Exclusion Criteria:

* Uncontrolled glaucoma
* Glaucoma requiring more than a single agent for IOP control
* Patients with a corneal thickness greater then 620 micrometers
* Female patients who are pregnant, nursing, or planning a pregnancy during the study
* Patient who has any situation or condition, which in the investigator's opinion, may put the patient at a significant risk, may confound the study result or may interfere significantly with the participation in the study
* Uncontrolled or labile hypertension
* At the conclusion of the washout period any study participant with an IOP lower than 22 or greater than 35 mmHg.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | Day one, every hour for twelve hours.
Heart Rate | Day one, every hour for twelve hours.
Blood Pressure | Day one, every hour for twelve hours.
Intraocular Pressure | Day two twice, once in the AM, once in the PM.
Intraocular Pressure | Day seven, once.
Intraocular Pressure | Day fourteen, once.
Intraocular Pressure | Day twenty one, once.
Intraocular Pressure | Day twenty eight, once.
Heart Rate | Day two twice, once in the AM, once in the PM.
Heart Rate | Day seven, once.
Heart Rate | Day fourteen, once.
Heart Rate | Day twenty one, once.
Heart Rate | Day twenty eight, once.
Blood Pressure | Day two twice, once in the AM, once in the PM.
Blood Pressure | Day seven, once.
Blood Pressure | Day fourteen, once.
Blood Pressure | Day twenty one, once.
Blood Pressure | Day twenty eight, once.

CONTACTS AND LOCATIONS:
Overall Officials: Padma Nanduri, MD, Principal Investigator; Michael Boone, MD, Study Director
Locations (1):
- Eye Surgical and Medical Associates, Visalia, California, United States